CLINICAL TRIAL: NCT05083364
Title: A Phase 1/2a Dose-Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and/or Pharmacodynamics of ARO-C3 in Adult Healthy Volunteers and in Adult Patients With Complement-Mediated Renal Disease
Brief Title: Study of ARO-C3 in Adult Healthy Volunteers and Patients With Complement Mediated Renal Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROC3-1001
Record Dates: First submitted 2021-10-08; First posted 2021-10-19 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: C3 Glomerulopathy; IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1, participants are randomized to receive either ARO-C3 or placebo. Participants,care providers, investigator and outcomes assessors are all blinded to treatment assignment. Part 2 in patients with C3G or IgAN is open-label and there is no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ARO-C3 (Healthy Volunteers) (Experimental): 1 or 2 doses of ARO-C3 by subcutaneous (sc) injection
  Interventions: Drug: ARO-C3
- Placebo (Healthy Volunteers) (Placebo Comparator): placebo calculated volume to match active treatment by sc injection
  Interventions: Drug: Placebo
- ARO-C3 (Adult Patients with C3G or IgAN) (Experimental): 3 doses of ARO-C3 by sc injection
  Interventions: Drug: ARO-C3

INTERVENTIONS:
Drug: ARO-C3 — ARO-C3 for sc injection
  Arms: ARO-C3 (Adult Patients with C3G or IgAN); ARO-C3 (Healthy Volunteers)
Drug: Placebo — sterile normal saline (0.9% NaCl) for sc injection
  Arms: Placebo (Healthy Volunteers)

SUMMARY:
The purpose of AROC3-1001 is to evaluate the safety, tolerability, pharmacokinetics and/or pharmacodynamics in adult healthy volunteers (HVs) and in adult patients with complement-mediated renal disease (C3 Glomerulopathy [C3G] and IgA Nephropathy [IgAN]). In Part 1 of the study, HVs will receive either one or two doses of ARO-C3 or placebo. In Part 2 of the study, adult patients with C3G/IgAN will receive 3 open-label doses of ARO-C3. Dose levels in Part 2 will be determined based on cumulative safety and pharmacodynamic data from Part 1.

ELIGIBILITY:
Inclusion Criteria (All Participants):

* Willing to provide written informed consent and to comply with study requirements
* Female participants must be non-pregnant/non-lactating
* Healthy volunteers must be willing to be vaccinated with a meningococcal and pneumococcal vaccine. C3G and IgAN participants must have been vaccinated or willing to undergo vaccination
* All participants must be willing to be vaccinated or have a history of vaccination for Haemophilus influenzae
* Body Mass Index (BMI) between 18.0 and 35.0 kg/m2
* 12-lead electrocardiogram (ECG) at Screening with no abnormalities that may compromise participant's safety at discretion of investigator
* Participants of childbearing potential must use highly effective contraception during the study and for at least 12 weeks following the end of the study or last dose of study drug, whichever is later. Males must not donate sperm during the study and for at least 12 weeks following the end of the study or last dose of study drug, whichever is later.
* No abnormal finding of clinical relevance at the Screening evaluation that, in the opinion of the investigator, could adversely impact participant safety or study results

Inclusion Criteria (C3G and IgAN Participants):

* Diagnosis of C3G or IgAN
* Clinical evidence of ongoing disease based on significant proteinuria
* Estimated glomerular filtration rate ≥30 mL/Min/1.73 m2 at Screening and currently not on dialysis
* Must be on a maximally recommended or tolerated dose of an angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB)

Exclusion Criteria (All Participants):

* Seropositive for human immunodeficiency virus (HIV) infection,hepatitis B virus, or hepatitis C virus
* History of recurrent or chronic infections
* Uncontrolled hypertension
* Regular use of alcohol within 30 days prior to Screening
* Use of illicit drugs within 1 year prior to Screening or positive urine drug screen at Screening
* History of meningococcal infection
* History of asplenia or splenectomy
* Known contraindication or history of anaphylactic reaction to any vaccine or vaccine component or prophylactic antibiotics planned for use in the study
* Any medical or surgical condition that, in the opinion of the investigator, would expose the participant to a significant safety risk or compromise the results of the study

Note: Additional Inclusion/Exclusion criteria may apply per protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and/or Serious Adverse Events (SAEs) at Day 169 | up to day 169 (End of Study [EOS])

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ARO-C3: Maximum Observed Plasma Concentration (Cmax) | up to 48 hours post-dose
PK of ARO-C3: Area under the Plasma Concentration Versus Time Curve from Zero to 24Hours (AUC0-24) | up to 48 hours post-dose
PK of ARO-C3: Area Under the Plasma Versus Time Concentration Curve from Zero to the Last Quantifiable Plasma Concentration (AUClast) | up to 48 hours post-dose
PK of ARO-C3: Area Under the Plasma Concentration Versus Time Curve from Zero Extrapolated to Infinity (AUCinf) PK of ARO-C3: | up to 48 hours post-dose
PK of ARO-C3: Terminal Elimination Half-Life (t1/2) | up to 48 hours post-dose
PK of ARO-C3: Apparent Total Body Clearance of ARO-C3 from Plasma (CL) | up to 48 hours post-dose
PK of ARO-C3: Volume of Distribution (Vz/F) | up to 48 hours post-dose

CONTACTS AND LOCATIONS:
Locations (16):
- Australia (3):
  - Research Site 1, Camperdown, New South Wales
  - Research Site 3, Concord, New South Wales
  - Research Site 2, Clayton, Victoria
- Research Site 2, Tbilisi, Georgia
- Germany (2):
  - Research Site 2, Cologne
  - Research Site 4, Erlangen
- Research Site, Auckland, New Zealand
- South Korea (6):
  - Research Site 1, Gamcheon, Busan
  - Research Site 2, Haeundae, Busan
  - Research Site 3, Daegu, Daegu
  - Research Site 4, Goyang-si, Gyeonggi-do
  - Research Site 6, Soeul
  - Research Site 8, Soeul
- Thailand (2):
  - Research Site 2, Bangkok
  - Research Site 3, Chiang Mai
- Research Site 4, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639